CLINICAL TRIAL: NCT02160964
Title: A Prospective Multi-center Study Using a Novel Algorithm to Improve the Retrieval Rate of Inferior Vena Cava Filters Placed Across the US
Brief Title: Using a Novel Algorithm to Improve the Retrieval Rate of Inferior Vena Cava Filters (iRetrieve Study)
Acronym: iRetrieve
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Heart and Vascular Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PC14-0610-002
Record Dates: First submitted 2014-06-07; First posted 2014-06-11 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Venous Thromboembolism,; Pulmonary Embolism,; Deep Vein Thrombosis,
Keywords: Inferior Vena Cava
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Since 2003, that the first retrievable IVC filter was introduced in the U.S,improvements have been made in the filter design to resolve problems of structural integrity and increase the ability to remove the filter after longer periods of time.The FDA issued a communication in August 2010 advising physicians to remove retrievable filters whenever possible and updated that letter again in May 2014 due to concerns that these retrievable IVC filters, intended for short-term placement, are not always removed once a patient's risk for PE subsides. Known long term risks associated with IVC filters include but are not limited to lower limb deep vein thrombosis (DVT), filter fracture, filter migration, filter embolization and IVC perforation.

DETAILED DESCRIPTION:
Several studies have shown that approximately 80% to 85% of optional IVC filters are never retrieved. The successful removal of retrievable filters requires diligent patient follow-up and interdepartmental cooperation, and even so, successful removal is not always possible. American College of Chest Physicians (ACCP) guidelines for IVCF placement indications advocates a close, structured follow-up of retrievable IVCFs to improve filter retrieval rates.

Using a retrieval algorithm and pathway program, a score will trigger a secure email and text messages sent to both physician and patient at different timelines, for follow up so as to retrieve filter placed.

ELIGIBILITY:
Inclusion Criteria:

* Data obtained in line with good clinical practice, applicable laws and regulation

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating study centers will enroll patients and enter data in the web-based platform that include demographics, clinical features, and clinical pathway
Sampling Method: Non-Probability Sample
Enrollment: 1786 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Filter retrieval rate | 24 Months

SECONDARY OUTCOMES:
Absence of major adverse event | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Uchenna Onyeachom, Study Director — Heart and Vascular Outcomes Research Institute; John Rectenwald, MD, Principal Investigator — University Of Michigan Health System, Ann Arbor